CLINICAL TRIAL: NCT05738785
Title: Risk of Osteoporotic Fracture in Home Care Patients in Turkey: A Call for Action
Brief Title: Risk of Osteoporotic Fracture in Home Care Patients in Turkey
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Uzm. Dr. Mustafa Hüseyin Temel, Uskudar State Hospital
Other Study IDs: 1
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis; Osteoporosis Risk; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home health care patients: Home health patients registered in the Anatolian side of Istanbul
  Interventions: Other: Document review and scanning

INTERVENTIONS:
Other: Document review and scanning — Osteoporosis risk and osteoporotic fracture risk will be calculated by examining the patients' files.

SUMMARY:
This study will assess the incidence of osteoporosis and osteoporotic fracture risk of registered home health patients in the Anatolian side of Istanbul.

DETAILED DESCRIPTION:
After selecting the patients who have been visited by the team in the last 6 months from the patients registered in the home health system, the number of patients required to reflect the population will be determined, and patient files will be selected by randomization. Demographic information, comorbidities, medications, and blood tests will be recorded. FRAX risks of the patients will be calculated, and it will be examined whether they have any previous fracture history and whether they have received treatment for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Being registered for home health services Having made a call to home health services in the last 6 months

Exclusion Criteria:

Patients that have passed away

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Home care patients who have called home health services in the last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
Osteoporotic fracture risk of home care patients | 3 months
  Osteoporotic fracture risk of home care patients

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar State Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No